CLINICAL TRIAL: NCT06125782
Title: Effect of Omega-3 Fatty Acid on Neurobehavioral Status of Children With Autism Spectrum Disorder: A Randomized, Double- Blind, Placebo Controlled Trial
Brief Title: Effect of Omega-3 Fatty Acid on Neurobehavioral Status of Children With Autism Spectrum Disorder: A Randomized, Double-Blind, Placebo Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Shawsun Tamanna Chowdhury, Effect of Omega-3 Fatty Acid on Neurobehavioral Status of Children with Autism Spectrum Disorder: A Randomized, Double-Blind, Placebo Controlled Trial, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: BSMMU/2023/5/965
Record Dates: First submitted 2023-07-05; First posted 2023-11-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 fatty acid (Active Comparator): One Omega-3 fatty acid softgel capsule 1 gm for children at or below 25 kg and two Omega-3 fatty acid softgel capsule above 25 kg. In this intervention arm having 32 participants, half will have plasma Omega 3 fatty acid level within reference value and rest half below reference value.
  Interventions: Drug: Omega 3 fatty acid
- Placebo (Placebo Comparator): Placebo softgels having almost same color and shape, one softgel for children at or above 25 kg and two softgels for children above 25 kg. In this placebo arm having 32 participants, half will have plasma Omega 3 fatty acid fatty acid level within reference value and rest half below reference value.
  Interventions: Drug: Placebo of Omega-3 fatty acid softgel capsule

INTERVENTIONS:
Drug: Omega 3 fatty acid — Omega 3 fatty acid 1 gm softgel capsule- 1 for children at or below 25 kg and two for above 25 kg.
  Arms: Omega-3 fatty acid
Drug: Placebo of Omega-3 fatty acid softgel capsule — Placebo of Omega-3 fatty acid softgel capsule- colour and shape almost similar to the original drug- 1 for children at or below 25 kg and 2 for above 25 kg.
  Arms: Placebo

SUMMARY:
This study is conducted to assess whether Omega-3 fatty acid improves neurobehavioral staus of children with Autism Spectrum Disorder and whether there is any correlation of this improvement with reference range of Omega-3 fatty acid.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a complex neurodevelopmental disorder of children with lifelong impacts. WHO estimates the international prevalence of ASD in 2022 at 1 in 100 children. Till date, no pharmacological treatment has been proven effective for ASD. This proposed study is an effort to explore whether Omega-3 fatty acid supplementation produces improvement in neurobehavioral symptoms of ASD. This study will be a randomized, double-blind, placebo-controlled trial.A total of sixty four (64) ASD patients attended in the outpatient department of IPNA, BSMMU will be selected for the study according to inclusion and exclusion criteria. Diagnosis of ASD will be made by DSM-V (Diagnostic and Statistical Manual of Mental Disorders, 5th edition). After completion of necessary formalities including informed consent of the patients, each participant will be assessed by translated and validated Bangla version of Aberrant Behaviour Checklist (ABC-parents rated). Omega-3 fatty acid ( Docosahexaenoic acid, DHA and Eicosapentaenoic acid, EPA) level in plasma will be measured in HPLC. 32 patients having DHA and EPA within reference value and 32 patients below the reference value will be selected. Then participants of each group will randomly be assigned into two groups: Intervention group and Control group. The intervention group patients will receive Omega-3 fatty acid 1 gm softgel once daily for 8 weeks at or below 25 kg and 1 gm softgel twice daily for 8 weeks above 25 kg making a total dose of 2gm/day. On the other hand, patients in control group will receive 1 placebo softgel of 1 gm once daily for 8 weeks at or below 25 kg and twice daily above 25 kg. After 8 weeks of therapy each participant will be assessed once again by Bangla version of ABC and plasma level of DHA and EPA will be measured.

ELIGIBILITY:
Inclusion Criteria:

Fulfills diagnosis of ASD by meeting DSM-5 diagnostic criteria. Written parental consent for participation. Age of children: 2-18 years. Sex: all.

-

Exclusion Criteria:

Those taking Omega-3 fatty acid or fish oil at present. Known allergy to fish or fish oil. Diagnosed with a psychotic disorder (e.g. Schizophrenia) or mood disorder, including depression or bipolar disorder.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Change of baseline ASD symptoms at 8 weeks evaluated by Aberrant Behavior Checklist(parent rated) | baseline and 8 weeks
  Change of ASD symptoms from baseline to 8 weeks measured by Aberrant Behavior Checklist (ABC)- community. ABC is a 58 item questionnaire designed to measure the symptoms of Autism spectrum disorder. It has 5 subscales- irritability, social withdrawal, stereotypic behavior, hyperactivity/ non-compliance, Inappropriate speech consisting of 15, 16, 7, 16 and 4 items respectively. The lower scores indicate better outcome.

SECONDARY OUTCOMES:
Change in baseline plasma DHA level at 8 weeks; Change in baseline plasma EPA level at 8 weeks. | baseline and 8 weeks
  Change in plasma DHA level from baseline to 8 weeks. Higher DHA level indicates better outcome.
Change in baseline plasma EPA level at 8 weeks; | baseline and 8 weeks.
  Change in plasma EPA level from baseline to 8 weeks. Higher EPA level indicates better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No